CLINICAL TRIAL: NCT01857596
Title: A Phase 1-b Non-blinded Study of Safety, Tolerability and Efficacy of Lorexys in Premenopausal Women With Hypoactive Sexual Desire Disorder
Brief Title: Phase 1b/2a Unblinded Study of Responses in Premenopausal Women With HSDD to Lorexys Evaluating Efficacy and Safety
Acronym: PURPLE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: S1 Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1P-104-1000
Record Dates: First submitted 2013-05-10; First posted 2013-05-20 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Hypoactive Sexual Desire Disorder (DSM-IV-TR Defined); Sexual Interest/Arousal Disorder (DSM-5 Defined)
Keywords: Female Sexual Dysfunction; Hypoactive Sexual Desire Disorder; Sexual Interest/Arousal Disorder; Lorexys; Premenopausal female health
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Bupropion; Trazodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupropion -> Lorexys LO -> Lorexys HI (Experimental): Crossover with all on positive comparator,lower-dose Lorexys,higher-dose Lorexys
  Interventions: Drug: bupropion, Lorexys low-dose, Lorexys moderate-dose

INTERVENTIONS:
Drug: bupropion, Lorexys low-dose, Lorexys moderate-dose — Lorexys is a proprietary fixed-dose combination of two agents
  Other Names: Lorexys is bupropion plus trazodone; Lorexys lower-dose is 225 mg per day.; Lorexys moderate-dose is 450 mg per day.

SUMMARY:
The purpose of this study is to investigate whether Lorexys is effective and safe to treat premenopausal women who have lost their sexual desire to a distressing degree.

DETAILED DESCRIPTION:
Women are diagnosed with Hypoactive sexual desire disorder (HSDD) if they experience chronic loss of desire for sex together with significant distress or interpersonal difficulties due to this lack of desire. HSDD can have a serious effect on emotional well-being and interpersonal relationships.

There are no U.S. Food and Drug Administration-approved treatments for HSDD. Off-label treatments include testosterone, which is not always effective and can be accompanied by side effects such as excess hair growth, acne, and decreases in high-density lipoprotein (HDL) cholesterol levels.

Research in laboratory animals and clinical observations in humans suggest that re-balancing chemical messengers in the brain may stimulate sexual desire. S1 Biopharma's Lorexys® is a novel use fixed-dose combination (FDC) in an oral pill. Lorexys® combines two agents intended to restore balance to the brain's centers that control sexual function. Such effects are hoped to help women with HSDD.

The compound is Phase 2-ready without prior trials (Phase I safety studies) because the two agents have often been used together; individually, they are FDA-approved for treating other disorders (depression, for example), and in a large US survey, the two were taken together in about 23% of patients who were prescribed one of the two agents.

This research study requires subjects to take three different study medications for four weeks each, with at least a one-week "wash-out" period after each, and to report on rating scales how they feel. The medication is open-label (the subjects can see which medication they are receiving). That should not interfere with the evaluations or cause a big "placebo effect" because only a low proportion of women with HSDD have responded to a placebo in prior research studies of other compounds when using the same measures of efficacy.

Participation lasts 16 weeks, with 8 clinic visits. A weekly, but no daily, self-rating is required between visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 to 50 and still having regular menstrual periods. Women with intact ovaries are classified as premenopausal for this study, even if they have had a hysterectomy. Women who have had both ovaries removed, even if under age 50 and with an intact uterus, are not acceptable for this study.
2. In a stable, monogamous, communicative, reasonably amicable relationship for at least one year
3. Meets DSM-IV-TR criteria for Generalized Acquired Hypoactive Sexual Desire Disorder and HSDD is her main sexual disorder
4. Over the prior month, didn't respond to sexual initiations by partner
5. At screen and baseline, low or no and infrequent or rare desire for sex
6. At screen, has clinically relevant sexual distress as per FSDS-R score
7. Otherwise healthy physically and mentally. Minor chronic conditions not affecting sexual function are allowed. Side effects from any continuing concomitant medications must be mild and stable or nil.
8. Not pregnant or lactating for six months; using medically reliable contraception, i.e., diaphragm or (male or female) condom and spermicide, IUD, tubal sterilization, hormonal contraception (oral, vaginal, or implant), or (if the investigator finds the patient credibly monogamous) vasectomy of male partner.
9. Gives informed consent for and is willing to undergo all of the scheduled evaluations
10. Prompt for screening and baseline visits, is cooperative, and takes reasonable directions without excessive explanations
11. Her sexual partner is in a monogamous relationship with her, is sexually unimpaired (erectile dysfunction allowed only if adequately treated), and is available to her at least half of the time (in days per week).

Exclusion Criteria:

1. Masturbates more than once a month.
2. Sexual aversion or sexual pain disorder
3. Chronic conditions that may reasonably be expected to be unstable or to affect sexual function (e.g., gastrointestinal bleeding, diabetes, frequent asthma, Major Depressive or anxiety disorder, history within the prior 6 months of suicidality or drug abuse; history of breast, cervical, uterine, ovarian or other systemic cancer).
4. BMI (a standard ratio of weight to height) over 35.0 (obese)
5. Requires CYP3A4, CYP 2B6, or CYP 2D6 strong inhibitor or inducer drugs
6. Takes any sex hormone other than an approved hormonal contraceptive
7. Takes an antiepileptic/mood stabilizer, antipsychotic, antidepressant, anti-anxiety, or hypnotic drug or has a history of allergic reaction to such drugs

9. Drinks more than 7 alcoholic drinks per week (12-oz beer, 4-oz wine, 1 ½ oz liquor etc) 10. Drinks more than 6 cups of coffee or tea per day 11. History of seizures 12. Long QT syndrome (QTc <=480 msec), other significant cardiovascular disease 13. moderate or severe dysfunction of the liver (any LFT >=3x ULN) or renal dysfunction (BUN > 30 or Cr >2.0) 14. Uses sedating antihistamines or prescription sedatives 15. History of blood clots or abnormal bleeding tendencies, including daily use of medications adversely affecting coagulation, e.g., NSAIDs, systemic corticosteroids, or >81 mg aspirin daily.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Desire domain of the Female Sexual Function Index | Four weeks after baseline
  One item asks how often the subject feels sexual desire, and another item asks how much she feels desire. One of five answers must be checked for each item.

SECONDARY OUTCOMES:
Change in Female Sexual Distress Scale-Revised | Four weeks after baseline
  The subject self-rates 13 negative feelings, such as frustration, bother, and unhappiness, that may have occurred because of her sexual problems.
Change in Side Effects Checklist - 24 item | 4 weeks after baseline
  The subject self-rates how much (if any) she has been bothered by each of the 24 symptoms that have been commonly reported with similar drugs, such as headache, sleepy, and anxious, from "not at all" to "extremely."
Patient's Global Impression of Change | 4 Weeks after baseline
  Subject self-rates how much, if any, her sexual disorder has changed since starting the current study medication (worse, same, or 4 degrees of improvement)
Change in blood pressure and pulse | Four weeks after baseline
  Blood pressure and pulse are taken lying and standing
Change in 12-lead electrocardiogram | 15 weeks (end of last treatment) after screen
  An electrocardiogram is used to measure the regularity of the heartbeat and how well electrical impulses are transmitted through the heart
Change in routine lab studies including pregnancy tests and screen for illicit drugs | Screen (wk 0), end of treatment/new baseline (wks 6, 11, 15)
  About two teaspoons of blood are drawn to measure blood cells and body chemistry, and to see if the patient has become pregnant or has taken unauthorized substances.

OTHER OUTCOMES:
Change in Columbia Suicide Severity Rating Scale, Screen Version (6 items) | 4 weeks after baseline
  Brief interview of 3-6 specified questions asking if the patient feels like, wants to, or plans to be dead

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Segraves, MD, PhD, Principal Investigator — Levine, Risen & Associates, Inc.; Molly Katz, MD, Principal Investigator — Katz and Kade, Inc.; Robert E Pyke, MD, PhD, Study Director — Chief Medical Officer, S1 Biopharma, Inc.
Locations (2):
- United States (2):
  - Robert Taylor Segraves, MD, PhD, Beachwood, Ohio
  - Molly Katz, MD, Cincinnati, Ohio

REFERENCES:
- [Background] Moll JL, Brown CS. The use of monoamine pharmacological agents in the treatment of sexual dysfunction: evidence in the literature. J Sex Med. 2011 Apr;8(4):956-70. doi: 10.1111/j.1743-6109.2010.02190.x. Epub 2011 Jan 27. PMID 21272265